CLINICAL TRIAL: NCT00531531
Title: Control and Prevention of Respiratory Infections in Cystic Fibrosis Patients: an Evaluation of the Emission Distance of P. Aeruginosa From the Respiratory Tract of Infected Persons Through Coughing and Conversation.
Brief Title: Evaluation of the Emission Distance of P. Aeruginosa From the Respiratory Tract of People With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: Italian Cystic Fibrosis Research Foundation (Other); Ospedale Meyer (Other)
Responsible Party: Principal Investigator, Filippo Festini, Associate Professor, University of Florence
Other Study IDs: FFC#16/2007
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Cystic Fibrosis
Keywords: pulmonary infection; transmission; P.Aeruginosa; surfaces
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
It is well known that an association exists between the acquisition of some respiratory pathogens and prognosis of CF people. About 57 % of patients has a lung infection due to P.aeruginosa (PA). Transmission of PA between CF patients is possible and several prevention measures are recommended. Among these measures, all international guidelines recommend that CF people maintain a minimum distance of 1 meter between them. However, this recommendation is not supported by specific studies and scientific evidence. In other words, the investigators don't know if this measure is sufficient or excessive, as it is based only on a theoretical rationale.

This study aims at measuring experimentally the distance that can be reached by PA emitted from airways of colonized CF patients during cough and during conversation.

To this purpose, the investigators will evacuate the presence of PA on surfaces placed at 4 different distances from patients, through the collection of 8 swabs, 4 of which following cough and 4 following conversation. Swabs will be collected on sterile surfaces comprised between tra 0 - 0,5 mt; 0,5 -1,00 mt.; 1,00 - 1,5 mt and 1.5-2 mt.

All the PA-positive CF patients of the CF Centre of Tuscany aged 14 or more will be recruited.

DETAILED DESCRIPTION:
Background

Cystic Fibrosis (CF) represents the most frequent genetic disorder with autosomal recessive transmission having a negative prognosis in Caucasian populations, with an incidence of about 1 in 3000. CF is a multisystemic disease involving the exocrine functions, in particular, of the respiratory tract and the gastroenteric system. The mutated gene causes an alteration in the transportation of chloride and sodium that leads to the production of denser bronchial secretion, favouring the onset of chronic respiratory infections, inflammations and respiratory insufficiency. Indeed, pulmonary infections are one of the primary characteristics, as well as the main cause of morbidity and mortality in CF.

There is an association between the acquisition of some respiratory pathogens (mainly B. cepacia complex [BCC] and P. aeruginosa [PA]) and the worsening of the parameters of respiratory function and a lower survival rate.

Recent epidemiological data show that 57.3% of CF patients have a pulmonary infection caused by PA.

Therefore, to prevent the clinical consequences deriving from chronic colonization of PA, avoiding contact with the infected patient when possible can be of fundamental importance.

The means by which the patient comes in contact with these pathogens is still not entirely clear; nevertheless, it is believed that transmission can occur through direct contact or droplets, or through indirect contact with inert surfaces used in common by colonized and non-colonized patients, or by reservoirs and surfaces in the care environment itself. Droplets are defined as large drops (>5 microns) produced by coughing, sneezing or speaking, or by the implementing of certain procedures such as aspiration or broncoscopy.

As for indirect means of transmission, it has been demonstrated that these pathogens have high survival rates on inert surfaces: for example, PA suspended in physiological solution can survive on dry surfaces for 24 hours and in patient expectoration for 8 days.

If expelled with coughing or sneezing from the CF patient's respiratory tract, therefore, PA and BCC [20] can linger on the surfaces of the health care centre for a long time, later to enter into contact with the respiratory mucosa of CF patients attending the same centre, through contact of the patients' hands on contaminated surfaces.

Only a limited number of studies has evaluated the prevalence of pathogens on non-critical surfaces in a CF centre.

In one recent study our research group evaluated over a 4-year period the prevalence of the pathogenic micro-organisms for CF in specimens taken from non-critical surfaces and sinks of an out-patient clinic dedicated exclusively to the care of CF patients, with the aim of improving the prevention of cross-infections in CF centres.

As for direct transmission of PA, there are various international prevention guidelines. All the guidelines include the recommendation that CF patients maintain a minimum distance of 1 meter between one another.

A recent study has demonstrated the theoretical possibility of airborne PA transmission.

Specific Aims and Rationale According to all international guidelines for controlling and preventing infections in CF patients, it is necessary to maintain a minimum distance of 1 meter from other CF patients in order to avoid the transmission of PA and BCC and the clinical consequences of a chronic infection from this pathogen. This indication derives from a similar recommendation contained in the CDC Guidelines on hospital isolation precautions relative to all infectious diseases transmitted through droplets. It is based on the theoretical assumption that, besides transmission by direct contact, the transmission of PA takes place prevalently through droplets.

There have been only two studies on the distance reached by PA emitted from the respiratory tract of CF patients. The first study [18] examined PA emission from CF patients' coughing, making them cough onto a dish held by the patients themselves, then onto a plate held at a distance of about a meter. In the second study six PA-colonized patients coughed in the direction of a soap bubble holder held at a distance of 10 cm, 20 cm, 30 cm, 40 cm and 50 cm from the mouth.

The results obtained in these two studies have shown the possibility of transmitting PA through coughing at a distance of at least one meter, and the possibility of emitting PA at distances greater than 40 cm. However, these studies do not provide proof that one meter is an effective indicator of the distance necessary for preventing PA emitted by one patient from reaching another.

It appears that no study has ever investigated if PA can be expelled from a carrier's respiratory tract by coughing at a distance greater than the recommended one meter "safety distance" between CF patients, and no study has been done on the maximum distance PA emitted during a normal conversation can reach.

In any case, aside from the distance PA can actually reach; there are no studies on the effectiveness of a 1-meter distance between CF patients as a measure for preventing PA cross-infections.

Since there are very few data available on how far PA emitted from the respiratory tract of a colonized CF patient through coughing can reach and no data relative to simple conversation, the recommendation of a one-meter distance does not seem to be backed up by sufficient evidence. In other words, one meter may not be a great enough distance for preventing the potential risk of transmission; therefore, the recommendation to maintain a minimum distance of one meter may be inadequate.

Our study thus intends to contribute to filling the knowledge gap to this regard, and to clarifying the validity of the minimum distance of one meter as a prevention measure in the transmission of PA from one CF patient to another.

The objectives in this study are:

* To evaluate what distance can be reached by PA expelled through the emission of droplets from the respiratory tract of a CF patient during a simple conversation and coughing.
* To verify if the 1-meter distance from patients colonized by PA is actually an effective prevention measure in regard to PA infection, as reported in the International Guidelines.

Experimental study not checked with convenience sample. This study will evaluate the distance reached by Pseudomonas aeruginosa after a normal conversation and after coughing by CF patients.

With this aim, we will evaluate the presence of PA on surfaces at 4 different distances from the patient, by culturing 8 swabs taken from the surfaces themselves, 4 of which after normal conversation and 4 others after coughing.

Data collection At the time of inclusion in the study the following data will be collected: Patient name and surname, age in months, Rx score, FEV1, BMI, Micro-organisms present in the previous and current expectorate culture, PCR.

After collecting the specimens and preparing the culture plates, PA growth in the mediums corresponding to the various collection distances will be observed.

The results of the laboratory analysis will be reported in the patient's file, thus:

Presence of Pseudomonas Aeruginosa

* after conversation: 0 - 0.5 m; 0.5 - 1.00 m; 1.00 - 1.5 m; 1.50 - 2.00 m.
* after coughing: 0 - 0.5 m; 0.5 - 1.00 m; 1.00 - 1.5 m; 1.50 - 2.00 m.

Safety measures Personnel will wear single-use gloves and coats.

Data management and statistical analysis The data will be entered into Microsoft Access 2000 database. For each of the four distances and for each of the two modes (coughing and conversation) the percentage of PA presence will be determined and the confidence intervals will be defined to 95% of the percentages.

Moreover, we will look for associations between the presence/absence of PA at each distance and for each of the modes, and the clinical variables in each patient.

For qualitative variables statistical analysis will be made with Chi-square test. For quantitative variables statistical analysis will be done with Student's T-distribution.

Expected Results:

We expect to obtain estimates of the proportion of contaminated areas so as to estimate the CF patient risk of being reached by secretions expelled from the respiratory tract of other CF patients at different distances.

Clinical protocols

Recruitment:

Upon a patient receiving a check-up at the CF Centre, the researcher will decide, on the basis of demographics and microbiology, if the patient can be included in the study group.

If the patient has reached the age of 14 and the last microbiological culture of his expectorate is positive for PA, the patient will be asked (and his parents, if under age) to participate in the study and will be given background information. After all his questions are answered, if the patient decides to participate his written consent will be taken (co-signed by his parents, if under age). Subsequently, the patient's entry data will be taken by filling out a patient questionnaire, after which the specimens will be collected.

The study does not call for the assignment of a therapeutic strategy; the clinical and laboratory data relative to the patients participating in the study will be obtained during routine follow-up, without modifying current clinical practice.

Specimen collection methods To collect the specimens, a special ruled table (0.5 X 2.10) will be set up and covered with a single-use waterproof surgical cloth after the patient has been enlisted in the study.

The patient will then be asked to place himself in front of the table at the 0 m point.

The table will be regulated according to the patient's height, at the level of his navel.

Then the patient will be asked to read a text placed in front of him out loud, in order to recreate a normal conversation.

We will then proceed to take the specimens with 4 sterile swabs, each one of which will be used for collecting specimens on the table surface subdivided into the following distances: 0 - 0.5 m; 0.5 - 1.00 m; 1.00 - 1.5 m; 1.50 - 2.00 m.

Specimen collection with a sterile swab from the surface of the sterile cloth will be done by rubbing entirely each of the four surfaces into which the sterile cloth is subdivided entirely, using a boustrophedonic movement.

After the first set is collected, the single-use cloth will be substituted in order to restore sterile conditions.

Next, the patient will be asked to perform two FET sequences which consist in giving one or two forced expirations with the glottis open, starting with medium-low lung volume, followed by a rest period in which diaphragm breathing is maintained. At this point the collection of the next 4 specimens will be taken in the method described above.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF
* Age 14 or older.
* PA infection documented by the most recent expectorate culture available, no more than 3 months old.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: People with CF attending the CF Center of Tuscany, aged 14 or older, with documented pulmonary Pseudomnas aeruginosa infection.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of surface samples positive for PA | six months

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Festini, BN, BSN, RN, Study Chair — University of Florence, Italy; Cesare Braggion, MD, Study Director — Cystic Fibrosis Center, Meyer Hospital Florence
Locations (1):
- Cystic Fibrosis Center of Tuscany, Meyer Hospital, Florence, Italy